CLINICAL TRIAL: NCT06472180
Title: Marginal Adaptation, Color Stability and Clinical Performance of Sectional and Full Glass Ceramic Laminate Veneers. A Randomized Clinical Trial
Brief Title: Sectional Versus Full Glass Ceramic Laminate Veneers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Nehal Gamal, Principal Investigator, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12
Record Dates: First submitted 2024-06-17; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Spacing of Anterior Teeth
Keywords: Mini-veneers; partial veneers; porcelain fragments; sectional veneers; laminate veneers

STUDY DESIGN:
Who Masked: Participant
Masking Description: double blinded Data analyst, statistician and patient will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention- Glass ceramic sectional veneer (Experimental): participants receive Glass ceramic sectional veneer covering only the area of defect
  Interventions: Procedure: Glass ceramic sectional veneer
- control-Glass ceramic laminate veneer (Active Comparator): participants receive laminate veneers made of glass ceramics as it is well documented in the literatures as successful restoration modality
  Interventions: Procedure: Glass ceramic laminate veneer

INTERVENTIONS:
Procedure: Glass ceramic sectional veneer — partial laminate veneer
  Arms: intervention- Glass ceramic sectional veneer
Procedure: Glass ceramic laminate veneer — Glass ceramic laminate veneer
  Arms: control-Glass ceramic laminate veneer

SUMMARY:
The aim of the study is to assess the marginal adaptation, color stability and clinical performance of glass ceramic sectional veneers compared to full laminate veneers There's two null hypotheses , the first is that there is no difference in the marginal adaptation of sectional and full glass ceramic laminate veneers.

the Second is that there is no apparent change in color stability and clinical performance of sectional and full glass ceramic laminate veneers.

DETAILED DESCRIPTION:
Although seeking for more minimally invasive treatment modalities with the use of the new advancements in ceramics and adhesive materials, however there is insufficient clinical studies assessing the ultraconservative sectional veneers has been published although there are many published case reports proving their success .

Hence the aim of this study is to assess the sectional veneers compared to laminate veneer regarding marginal adaptation, color stability and clinical performance

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking for esthetics with the following criteria
* Male or female patients age range above 18 years old
* Minor esthetic defects in anterior region
* Multiple spacing
* diastemas
* Incisal fracture
* Initial proximal caries
* Patients able physically and psychologically to tolerate restorative procedures
* Patients willing to return for follow-up examinations and evaluation
* Class I occlusion

Exclusion Criteria:

* Patients free of:
* Tempromandibular disorders
* Para-functional habits
* Cracked teeth
* Moderate or deep caries
* Heavily discolored teeth
* Heavy smokers
* Enamel defects compromising bonding
* Active periodontal disease
* Pulpal disease
* Mobility
* Occlusal disturbances
* Class II and III occlusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation of sectional and full glass ceramic laminate veneer using digital device intraoral scanner | Baseline,3,6,9,12 months
  assessment of the marginal adaptation using digital device intraoral scanner software

SECONDARY OUTCOMES:
Color stability | Baseline,3,6,9,12 months
  assessment of the Color stability using intraoral scanner
Clinical performance | Baseline,3,6,9,12 months
  categorical outcome of clinical performance using FDI(World Dental Federation) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Nehal G Mohamed, BDS, Principal Investigator — October University for Modern Sciences & Arts
Locations (1):
- October University for Modern Sciences & Arts, Giza, Giza, 6th October City, Egypt

IPD SHARING:
Plan to Share IPD: Undecided